CLINICAL TRIAL: NCT02166151
Title: Efficacy and Safety of Omalizumab in Chronic Idiopathic Urticaria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Michael David, Prof. Michael David, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0550-31 -RMC
Record Dates: First submitted 2014-05-28; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omalizumab (Experimental): Omalizimab 150 mg S.C. once a month for consecutive 3 months
  Interventions: Drug: Omalizimab

INTERVENTIONS:
Drug: Omalizimab — Omalizimab 150 mg S.C. once a month for consecutive 3 months
  Other Names: Xolair

SUMMARY:
The study is designed to assess the efficacy and safety of monthly injections of Omalizumab 150 mg for 3 consecutive months, in patients with chronic idiopathic urticaria, unresponsive to convetional therapy by antihistamins or oral corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic idiopathic urticaria for 3 months
* failure on treatment with at least 2 antihistamins and systemic corticosteroids or cyclosporin

Exclusion Criteria:

* physical or cholinergic urticaria
* past treatment in Omalizumab i nprevious year
* parasitic infection
* malignancy in last 5 years
* known sensitivity to Omalizumab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with ≥ 50% Decrease in Urticaria Activity Score (UAS) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael David, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel, Israel